CLINICAL TRIAL: NCT07304011
Title: A Phase 2 Study of Olutasidenib in Combination With Azacitidine Followed by Olutasidenib Maintenance After Venetoclax Plus a Hypomethylating Agent Regimen (HMA-VEN) for IDH1-Mutated Acute Myeloid Leukemia (AML)
Brief Title: Olutasidenib With Azacitidine Followed by Olutasidenib Maintenance for the Treatment of IDH1-mutated Acute Myeloid Leukemia in Patients With Prior Treatment With Venetoclax Plus a Hypomethylating Agent
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC320; NCI-2025-09023 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC320 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2025-12-23; First posted 2025-12-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; olutasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (olutasidenib, azacitidine) (Experimental): Patients receive olutasidenib PO BID on days 1-28 of each cycle and azacitidine IV or SC for seven days of each cycle as per schedule determined by investigator. Cycles repeat every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive olutasidenib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and biopsy and blood sample collection throughout the study.
  Interventions: Drug: Azacitidine; Drug: Olutasidenib

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Olutasidenib — Given PO
  Other Names: FT 2102; FT-2102; FT2102; IDH1-R132 Inhibitor FT-2102; Rezlidhia

SUMMARY:
This phase II trial studies how well giving olutasidenib with azacitidine, followed by olutasidenib maintenance, works in treating patients with IDH1-mutated acute myeloid leukemia (AML) who have received prior treatment with venetoclax plus a hypomethylating agent (HMA-Ven). Olutasidenib and azacitidine may inhibit the growth of cancer cells by blocking certain enzymes required for cell growth. Maintenance therapy can help prevent or delay cancer from coming back. Olutasidenib with azacitidine followed by olutasidenib maintenance may be effective in treating patients with IDH1-mutated AML who have received prior HMA-Ven.

DETAILED DESCRIPTION:
Participants receive olutasidenib orally (PO) twice daily (BID) on days 1-28 of each cycle and azacitidine intravenously (IV) or subcutaneously (SC) for seven days of each cycle as per schedule determined by the investigator. Cycles repeat every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive olutasidenib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and biopsy, and blood sample collection throughout the study.

After completion of study treatment, patients are followed up within 30 days and then every 4 months until withdrawal of consent, lost to follow-up, study termination, or death.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented AML (except acute promyelocytic leukemia with the t(15;17) translocation) as defined by the World Health Organization (WHO) or International Consensus Classification criteria
* Achieved complete response (CR)/complete remission with incomplete count recovery (CRi) response to first line HMA-Ven according to the European Leukemia Net (ELN) recommendations for diagnosis as determined by investigator review
* Documented IDH1-R132 mutations (≥ 0.01%) detected in the bone marrow or blood. Mutation must be present at the time of AML diagnosis or after initiating HMA-Ven
* Receiving first-line HMA-Ven with less than or equal to 4 cycles of HMA-Ven at the time of enrollment. Participants must discontinue venetoclax (Ven) at least 1 week (or 5 half-lives, whichever is shorter) from initiating study treatment
* Candidate for standard of care azacitidine
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 50%)
* No prior solid organ allograft
* Recovery from the non-hematologic toxic effects of prior treatment to grade ≤ 1, or baseline value according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) classification (excluding infertility or alopecia)
* Aged ≥ 18 at the time of consent
* Creatinine clearance ≥ 40 mL/min (calculated by the Cockcroft-Gault formula or measured by 24-hour urine collection)
* Serum alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN)
* Serum aspartate aminotransferase (AST) ≤ 3 × ULN
* Bilirubin ≤ 2 x ULN unless due to Gilbert's syndrome or controlled autoimmune hemolytic anemia (not requiring immunosuppressive other than ≤ 20 mg of prednisolone daily)

  * Note: Patients with Gilbert's syndrome may be included if total bilirubin is ≤ 3 × ULN and direct bilirubin is ≤ 2 × ULN
* Prothrombin time (PT) or international normalized ratio (INR)/activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN
* Women of child-bearing potential, men, and their respective partners, must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days after the last dose of olutasidenib
* Must sign and date the informed consent form prior to undergoing any study procedures

Exclusion Criteria:

* Prior IDH1 inhibitor (IDH1i) targeted therapy
* Prior AML therapy except for HMA-Ven
* History of a different malignancy unless they have been disease-free for at least 12 months and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with a history of other malignancies within 12 months and without any evidence of disease progression or requiring therapy may be considered, but only after consideration and approval by the Overall Principal Investigator (PI). Individuals with the following cancers are eligible if diagnosed and/or treated within the past 12 months: cervical cancer in situ, breast ductal carcinoma in situ (DCIS), and basal cell or squamous cell carcinoma of the skin
* Patients with symptomatic central nervous system (CNS) metastases or other tumor location (such as spinal cord compression, other compressive mass, uncontrolled painful lesion, bone fracture, etc.) necessitating an urgent therapeutic intervention, palliative care, surgery or radiation therapy
* Patients with previous allogeneic hematopoietic stem cell transplantation (HSCT) for non-AML indications, if they meet any of the following criteria: < 100 days from time of HSCT; active acute or chronic graft versus (vs.) host disease (GvHD); or receiving immunosuppressive therapy as treatment or prophylaxis against GvHD

  * Note: Doses < 20 mg methylprednisolone (or its equivalent) daily are not an exclusion criterion
* Treatment with radiation therapy or major surgery (requiring general anesthesia) within 2 weeks prior to study drug dosing
* Patients unable to swallow oral medications, or patients with gastrointestinal conditions (e.g., malabsorption, resection, etc.) deemed by the Investigator to jeopardize intestinal absorption
* Congestive heart failure (New York Heart Association Class III or IV) or unstable angina pectoris; previous history of myocardial infarction within one year prior to study entry, uncontrolled hypertension, or uncontrolled arrhythmias
* Patients with a baseline corrected QT interval by Fridericia's formula (QTcF) of > 480 msec

  * Note: This criterion does not apply to patients with a bundle branch block (BBB); for participants with BBB, a cardiology consult is recommended to ensure that QTcF is not prolonged
* Concomitant medication(s) known to cause Torsades de Pointes (TdP) initiated less than the duration required to reach steady-state plasma concentration (approximately five half-lives) before first dose of study drug. Medications used as needed (PRN), e.g. Zofran, and common AML supportive care drugs (e.g. levofloxacin, azoles, etc.) are exempt
* Concurrent treatment with chronic corticosteroids except if chronic treatment with < 20 mg of methylprednisolone daily or equivalent (pulse steroids for treatment or prophylaxis are allowed [e.g., for transfusion or medication reactions])
* Known history of seropositivity for HIV infection
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy (prophylactic systemic antimicrobials permitted)
* Uncontrolled disease-related metabolic disorder (e.g., hypercalcemia)
* Pregnant, breastfeeding, or planning to become pregnant while enrolled in this trial or within 90 days after the last dose of olutasidenib. Pregnant or breastfeeding

  * NOTE: Breast milk cannot be stored for future use while the mother is being treated on study)
* Plans to donate sperm or conceive a child through intercourse while enrolled in this trial or within 90 days after the last dose of olutasidenib
* Unwillingness or inability to comply with procedures either required in this protocol or considered standard of care
* Medical, uncontrolled disease-related metabolic disorder, psychiatric, cognitive, or other conditions that may, in the opinion of the investigator, compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol, or complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2031-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | At 12 months from complete response (CR)/complete remission with incomplete count recovery (CRi)
  Defined as the percent of patients who reached death due to acute myeloid leukemia (AML), relapse, or discontinuation of treatment due to an adverse event, at 12 months from the time of CR/CRi in patients with AML who begin first line venetoclax plus a hypomethylating agent regimen and subsequently transition to olutasidenib maintenance. The Kaplan-Meier method will be employed to summarize the duration from the initiation of study treatment to treatment failure and to report the probability of being event-free at one year. The 1-year treatment failure rate will be reported along with its 95% confidence interval.
Median time to treatment failure | From CR/CRi through death due to AML, relapse, or treatment discontinuation due to adverse event, assessed up to 4 years
  Will be reported along with its 95% confidence interval.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after last dose of study drug
  All AEs will be listed, documenting the course, outcome, severity, and relationship to the study treatment. The proportion of participants experiencing AEs, serious adverse events, and treatment delays will be reported. Incidence rates of AEs and the proportion of participants prematurely withdrawn from the study due to AEs will be reported. AEs will be classified by severity and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Relapse free survival | From the date of remission until the occurrence of hematologic relapse or death from any cause, assessed up to 4 years
  Relapse categorized as CR, complete remission with partial hematologic recovery (CRh), or CRi, will be determined according to the European Leukemia Net (ELN) guidelines. Will be summarized using the Kaplan-Meier method. Will be reported along with its 95% confidence interval.
Duration of remission | From the achievement of remission to hematologic relapse or death due to AML, assessed up to 4 years
  Remission categorized as CR, CRh, or CRi, will be determined according to the ELN guidelines. Will be summarized using the Kaplan-Meier method. Will be reported along with its 95% confidence interval.
Overall survival | From remission until death due to any cause, assessed up to 4 years
  Will be summarized using the Kaplan-Meier method. Will be reported along with its 95% confidence interval.
Rate of allogeneic hematopoietic cell transplants | Up to 4 years
  The proportion of patients receiving allogeneic hematopoietic cell transplants during the study period will be reported, along with its 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Jonas, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States